CLINICAL TRIAL: NCT05052606
Title: INSIGHTS Registry - Inspiring New Science In Guiding Healthcare in Turner Syndrome
Brief Title: Inspiring New Science In Guiding Healthcare in Turner Syndrome Registry
Acronym: INSIGHTS
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 19-3027
Record Dates: First submitted 2021-08-20; First posted 2021-09-22 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — If resources are available and optional consent is provided, a 5-10mL blood sample will be obtained in 1 gold top and 1 purple top (EDTA) tube and processed for storage of plasma, serum, and buffy coat. These specimens will be stored in a biobank with a barcode to link the sample with the patient for future studies involving the assessment of hormones, proteins, metabolites, DNA, RNA, and other studies. Phlebotomy will be combined with clinical phlebotomy whenever possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This study is an observational study without treatment intervention.

SUMMARY:
INSIGHTS is a registry research study that collects key information on medical history for girls and women with Turner syndrome and the clinical care they receive. This includes genetic tests, imaging, medications, and more for hundreds of patients seen at a number of clinics across the US. In addition to learning a lot about the current state of health for individuals with TS, INSIGHTS serves as an infrastructure to conduct future studies are meaningful to patients and their families.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with TS and TS variants as defined by the TS Clinical Practice Guideline definition (karyotype consistent with TS, phenotypic female, clinical feature(s) of TS)
2. Informed consent/assent as appropriate

Exclusion Criteria:

a. Lack of a TS diagnosis on file

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population for this registry is patients diagnosed with Turner syndrome who are seen at a participating clinic.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Health conditions | From study start until condition observed, up to 15 years
  Average number of chronic diagnoses per person

SECONDARY OUTCOMES:
Prevalence of mental health diagnoses | From study start until condition observed, up to 15 years
  Prevalence of mental health diagnoses is defined as the number of participants in the sample diagnosed with a mental health disorder by a clinician according to their medical record out of the total sample. This will be determined by a diagnosis of any of the following in a clinical encounter, problem list, and/or past medical history:
  * Depression
  * Anxiety
  * Mood disorder NOS
  * Psychotic disorder
  * Attention-deficit/hyperactivity disorder (ADHD)
  * Autistic disorder
Prevalence of premature ovarian insufficiency | From study start until condition observed, up to 15 years
  Prevalence of premature ovarian insufficiency is defined as the number of participants in the sample with a diagnosis of premature ovarian insufficiency (or failure) in their medical record clinical encounter, problem list, and/or past medical history or laboratory results in their medical record consistent with this diagnosis (elevated FSH or undetectable AMH) out of the total sample.
Prevalence of hearing loss | From study start until condition observed, up to 15 years
  Prevalence of hearing loss is defined as the number of participants in the sample formally diagnosed with a hearing loss in their medical record in a clinical encounter, problem list, and/or past medical history or an audiology report consistent with hearing impairment out of the total sample.
Cardiometabolic diagnoses - prevalence of obesity | From study start until condition observed, up to 15 years
  Prevalence of obesity is defined as the number of participants in the sample with obesity in their medical record out of the total sample. Obesity in pediatric populations is determined using BMI-for-age and obesity in adult populations is determined using BMI. BMI is calculated as the weight in kilograms divided by the height in meters squared.
  Participants will be considered to have obesity if:
  * There is a diagnosis of obesity in the medical record in a clinical encounter, problem list, and/or past medical history
  * For children 17 years and younger: there is an available growth chart/height/weight/other data necessary to calculate the BMI-for-age and the BMI-for-age is at or above the 95th percentile
  * For adults 18 years and older: there is a BMI at or above 30 kg/m2 or the data necessary to calculate BMI and it is at or above 30 kg/m2
Cardiometabolic diagnoses - prevalence of dyslipidemia | From study start until condition observed, up to 15 years
  Prevalence of metabolic syndrome is defined as the number of participants in the sample with dyslipidemia in their medical record out of the total sample. Dyslipidemia will be defined as:
  * Diagnosis of dyslipidemia, hypertriglyceridemia, hypercholesterolemia in a clinical encounter, problem list, and/or past medical history
  * Laboratory evidence of elevated total cholesterol, LDL, triglycerides, and/or low HDL for sex and age
Cardiometabolic diagnoses - prevalence of fatty liver disease | From study start until condition observed, up to 15 years
  Prevalence of fatty liver disease is defined as the number of participants in the sample with a formal diagnosis of fatty liver disease in their medical record out of the total sample. Fatty liver disease diagnosis in the medical record in a clinical encounter, problem list, and/or past medical history may also present as:
  * Non-alcoholic fatty liver disease (NAFLD)
  * Hepatic steatosis
  * Simple fatty liver disease
  * Non-alcoholic steatohepatitis
Cardiometabolic diagnoses - prevalence of hypertension | From study start until condition observed, up to 15 years
  Prevalence of hypertension is defined as the number of participants in the sample with evidence of hypertension in their medical record out of the total sample. Evidence of hypertension includes:
  * Formal diagnosis of hypertension in a clinical encounter, problem list, and/or past medical history
  * For children under 13 years old: a blood pressure reading at or above the 95th percentile for age, height, and sex
  * For children between 13 and 17 years old: a blood pressure reading at or above 130/80 mmHg
  * For adults 18 years or older: a blood pressure reading at or above 140/90 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Shanlee M Davis, MD, PhD, Principal Investigator — Children's Hospital Colorado
Locations (10):
- United States (10):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National, Washington D.C., District of Columbia
  - Lurie Children's, Glenview, Illinois
  - University of Kansas, Lawrence, Kansas
  - UNC Hospitals Children's Specialty Clinic, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Childern's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Seattle Children's, Seattle, Washington